CLINICAL TRIAL: NCT06393127
Title: Bioequivalence of the BI 1015550 High Dose Formulation C2 and the BI 1015550 High Dose Formulation C1 (Phase 3 Formulation) Following Oral Administration in Healthy Subjects (an Open-label, Randomised, Single-dose, Two-way Crossover Trial)
Brief Title: A Study in Healthy People to Compare How 2 Different High Dose Formulations of BI 1015550 Are Taken up in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0037; 2023-509950-67-00 (Registry Identifier: CTIS); U1111-1301-0834 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test treatment (T), then reference treatment (R): T-R (Experimental): Healthy subjects were administered one tablet of nerandomilast (Formulation C2) (Test treatment - T). After a washout period of at least 10 days, subjects were administered one tablet of nerandomilast (Formulation C1 - phase 3 formulation) (Reference treatment - R).
  Both treatments were administered orally with approximately 240 milliliters (mL) of water after an overnight fast of at least 10 hours (h). After drug administration, subjects additionally fasted for 4 h.
  Interventions: Drug: Nerandomilast
- Reference treatment (R), then test treatment (T): R-T (Experimental): Healthy subjects were administered one tablet of nerandomilast (Formulation C1 - phase 3 formulation) (Reference treatment - R). After a washout period of at least 10 days, subjects were administered one tablet of nerandomilast (Formulation C2) (Test treatment - T).
  Both treatments were administered orally with approximately 240 mL of water after an overnight fast of at least 10 h. After drug administration, subjects additionally fasted for 4 h.
  Interventions: Drug: Nerandomilast

INTERVENTIONS:
Drug: Nerandomilast — One dose of Formulation C2 (Test treatment - T) administered with approximately 240 mL of water after an overnight fast of at least 10 h. After drug administration, subjects additionally fasted for 4 h.
  Other Names: BI 1015550; JASCAYD®
Drug: Nerandomilast — One dose of Formulation C1 - phase 3 formulation (Reference treatment - R) administered with approximately 240 mL of water after an overnight fast of at least 10 h. After drug administration, subjects additionally fasted for 4 h.
  Other Names: BI 1015550; JASCAYD®

SUMMARY:
The main objective of this trial is to establish the bioequivalence of the BI 1015550 Formulation C2 (Test, T) and the BI 1015550 Formulation C1 (Reference, R), following a single oral dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subject according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 50 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial Further inclusion criteria apply.

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm) at screening
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin) or renal parameters (creatinine) exceeding the upper limit of normal (ULN) at screening
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a open-label, randomised, single-dose, two-way crossover trial in healthy subjects to compare the test treatment (T - nerandomilast [BI 1015550] Formulation C2) to the reference treatment (R - nerandomilast Formulation C1, as the phase 3 formulation). Subjects were randomly allocated to the 2 treatment sequences (T-R or R-T), and there was a washout period of at least 10 days between the administration of each treatment.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Screening procedures also included physical examination, check of vital signs, electrocardiogram, safety laboratory, demographics, relevant medical history, concomitant therapy. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Treatment period 1
Arm/Group | Test treatment (T), then reference treatment (R): T-R | Reference treatment (R), then test treatment (T): R-T
Started | 32 | 32
Completed | 32 (One subject received the wrong treatment.) | 32 (Three subjects received the wrong treatment.)
Not Completed | 0 | 0
Period: Washout period
Arm/Group | Test treatment (T), then reference treatment (R): T-R | Reference treatment (R), then test treatment (T): R-T
Started | 32 | 32
Completed | 30 | 32
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Non-compliance from subject with trial procedures | 1 | 0
Period: Treatment period 2
Arm/Group | Test treatment (T), then reference treatment (R): T-R | Reference treatment (R), then test treatment (T): R-T
Started | 30 | 32
Completed | 30 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): includes all subjects who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Treatment (T), Then Reference Treatment (R): T-R | Reference Treatment (R), Then Test Treatment (T): R-T | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (8.4) | 35.0 (8.3) | 35.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 15 | 18 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 29 | 32 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 28 | 32 | 60
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of nerandomilast (R-BI 1015550) in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: "subjects within sequences" as random effect, "sequence", "period" and "treatment" as fixed effects. These quantities were then back-transformed to the original scale.
Time Frame: Within 3 h prior to drug administration, and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 34, 48, 58, 72, 96, 120, 144 h after drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): includes all subjects in the TS who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if they contributed only 1 PK parameter value for 1 period to the statistical assessment. Only participants with available PK data are included in the analysis.
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/Liter (h*nmol/L)
Groups:
- Test treatment (T): Healthy subjects were administered one tablet of nerandomilast (Formulation C2) orally with approximately 240 mL of water after an overnight fast of at least 10 h. After drug administration, subjects additionally fasted for 4 h.
- Reference treatment (R): Healthy subjects were administered one tablet of nerandomilast (Formulation C1 - phase 3 formulation) orally with approximately 240 mL of water after an overnight fast of at least 10 h. After drug administration, subjects additionally fasted for 4 h.
Arm/Group | Test treatment (T) | Reference treatment (R)
Number analyzed (Participants) | 63 | 57
hour*nanomole/Liter (h*nmol/L) | 2275.77 (NA) — Adjusted geometric standard error = 1.04 | 2166.70 (NA) — Adjusted geometric standard error = 1.05
Statistical Analysis 1: Comparison: Test treatment (T) vs Reference treatment (R); Ratio of adjusted geometric means was calculated using an analysis of variance (ANOVA) model on the logarithmic scale. PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: "subjects within sequences" as random effect, "sequence", "period" and "treatment" as fixed effects. These quantities were then back-transformed to the original scale; Test type: Other; Ratio of adjusted geometric means [%] = 105.03, 90% CI 2-sided [99.07 to 111.36] — Ratio [%] = (adjusted geometric mean of T / adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 18.8

2. Primary Outcome: Maximum Measured Concentration of Nerandomilast in Plasma (Cmax)
Description: Maximum measured concentration of nerandomilast (R-BI 1015550) in plasma (Cmax) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: "subjects within sequences" as random effect, "sequence", "period" and "treatment" as fixed effects. These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) parameter analysis set (PKS): includes all subjects in the TS who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if they contributed only 1 PK parameter value for 1 period to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | Test treatment (T) | Reference treatment (R)
Number analyzed (Participants) | 63 | 58
nanomole/Liter (nmol/L) | 417.47 (NA) — Adjusted geometric standard error = 1.05 | 368.38 (NA) — Adjusted geometric standard error = 1.06
Statistical Analysis 1: Comparison: Test treatment (T) vs Reference treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 113.32, 90% CI 2-sided [102.70 to 125.05] — Ratio [%] = (adjusted geometric mean of T / adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 32.8

3. Secondary Outcome: Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of nerandomilast (R-BI 1015550) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
  Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model, which included effects accounting for the following sources of variation: "subjects within sequences" as random effect, "sequence", "period" and "treatment" as fixed effects. These quantities were then back-transformed to the original scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hour*nanomole/Liter (h*nmol/L)
Arm/Group | Test treatment (T) | Reference treatment (R)
Number analyzed (Participants) | 63 | 57
hour*nanomole/Liter (h*nmol/L) | 2298.06 (NA) — Adjusted geometric standard error = 1.04 | 2189.77 (NA) — Adjusted geometric standard error = 1.04
Statistical Analysis 1: Comparison: Test treatment (T) vs Reference treatment (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means [%] = 104.95, 90% CI 2-sided [99.10 to 111.14] — Ratio [%] = (adjusted geometric mean of T / adjusted geometric mean R)*100. Intra-individual geometric coefficient of variation (gCV) [%] = 18.5

ADVERSE EVENTS:
Time Frame: Adverse events: from drug administration up to 7 days. All-cause mortality: from drug administration until end of study examination, up to 37 days.
Description: Treated set (TS): includes all subjects who were treated with at least one dose of trial drug.
Arm/Group | Reference treatment (R) | Test treatment (T)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/63
Other Adverse Events (participants affected / at risk) | 5/59 | 2/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reference treatment (R) (N=59) | Test treatment (T) (N=63)
Headache (Nervous system disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT06393127/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT06393127/SAP_001.pdf